CLINICAL TRIAL: NCT06373874
Title: The Effect of High Reality Simulation Environment on the Skills of Midwifery Students, Learning Satisfaction, Anxiety and Self-Efficacy in Newborn Heel Blood Collection
Brief Title: The Effect of High Reality Simulation Environment on the Skills of Midwifery Students, in Newborn Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Yonca Çiçek Okuyan, Celal Bayar University, Midwifery Department, Research Assistant Dr., Manisa Celal Bayar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCBU-SBF-YC-04
Record Dates: First submitted 2024-04-08; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Students; Educational Problems; Anxiety
Keywords: Skills training; high reality simulation environment; skills laboratory; midwifery training.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment experimental study with experimental and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: group that practices in a high-reality simulation environment (Experimental): The researcher showed the student how to take heel blood on the model. The researcher introduced both high-reality simulation environment. As a pre-test, the student was asked to fill out the Introductory Information Form, Self-Efficacy-Efficacy Scale and State and Trait Anxiety Scales surveys. Midwifery students in the experimental group were asked to take heel blood on a model in a high-reality simulation environment.Heel blood collection skill evaluation form was filled out by the researcher.As a post-test, the student was asked to fill out the Introductory Information Form, Self-Efficacy Scale and State and Trait Anxiety Scales surveys.
  Interventions: Behavioral: Heel blood collection in a newborn simulation model
- control group (No Intervention): They took heel blood on a newborn model in the simulation room as routine training.

INTERVENTIONS:
Behavioral: Heel blood collection in a newborn simulation model — The person who will take heel blood in the newborn simulation model can prepare the materials.
  Firstly, the blood sample can fill in all the information on the filter paper. Knows where the baby's face should be. It can determine the area where a heel blood sample can be taken.It can gently warm the heel area for a few minutes. The area can be cleaned with alcoholic preparation (cotton/swab, etc.). He can squeeze the heel with his thumb and index finger in front. The other 3 fingers can be rubbed at the back. May stroke the heel three times. The heel can be pierced once with a lancet at a suitable location. He can relax his hand. He can wipe away the first drop of blood. It can create a large thick drop of blood to be collected on filter paper. It can make the drop fill the entire ring on the filter paper with one touch. After the procedure is completed, the heel can be pressed.
  Arms: Experimental: group that practices in a high-reality simulation environment

SUMMARY:
The researchers gave midwifery students theoretical training on how to take heel blood on a newborn model. Students were asked to take heel blood on the model in the high-reality simulation environment and simulation room. The student's ability to take heel blood before and after taking heel blood in a high-reality simulation environment or on a newborn model in a simulation environment, satisfaction with learning, anxiety and self-efficacy levels were compared.

DETAILED DESCRIPTION:
The population of the research consisted of 4th grade midwifery students studying in the fall semester of the 2022-2023 academic year (N = 98). 6 students could not continue studying. No sample selection was made and an attempt was made to reach the entire universe. The sample of the research consisted of a total of 92 midwifery students, n=46 in the control group and n=46 in the experimental group. Verbal and written permission was obtained from the students included in the research. Both the experimental and control groups were given theoretical training on heel blood collection on a model using the show-and-tell technique.Then, those in the experimental group were asked to take heel blood on a newborn model in a high-reality simulation environment. The control group was asked to take heel blood on a newborn model in the simulation laboratory. Self-Efficacy-Efficacy scale for both the experimental group and the control group. State and Trait Anxiety Scale was applied as pre-test and post-test. Student Satisfaction and Self-Confidence in Learning Scale was applied only as a posttest. The heel prick skill evaluation form was filled out by a researcher. Pre-test and post-test results, Student tudent Satisfaction and Self-Confidence in Learning scores , and Heel Blood Skill scores were compared between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade students (n=49) who took the Maternal and Child Health Practice course of the Midwifery Department and agreed to participate in the study voluntarily were included in the study.

Exclusion Criteria:

* Students in younger grades who did not take the Maternal and Child Health Practice course were excluded.

Ages: 21 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Midwifery students
Enrollment: 92 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Skill checklist | during the intervention
  The heel prick skill (20 tasks/step) is based on checklists for evaluating student management, recommendations of the Ministry of Health and WHO, and training materials and guides prepared by the Ministry of Health. Each task/step was evaluated as "outstanding" if performed completely and correctly, and as "needs improvement" if performed incompletely and incorrectly. Needs improvement is rated as 1 point, sufficient as 2 points. As a result of the skill checklist, the lowest score is 1 and the highest score is 40
State and Trait Anxiety Scales | one hour before and one hour after interventions
  It is used to determine state and trait anxiety levels in individuals. State-Trait Anxiety Scale consists of a total of 40 items, 20 items each. The State Anxiety Scale requires the individual to describe how he or she feels at a particular moment and under certain circumstances. The total score of the scale varies between 20-80. A high score from the scale indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Self-Efficacy Scale | one hour before and one hour after interventions
  The scale was developed to determine behavior and behavioral changes. The scale consisting of 23 items is a 5-point Likert type self-evaluation scale. It includes the options 1-"does not describe me at all", 2-"describes me a little", 3-"undecided", 4-"describes me well", 5-"describes me very well" and the score given for each item is taken as basis. Scores between 23 and 115 are obtained from the scale. A minimum of 23 and a maximum of 115 points can be obtained from the entire scale. A high total score from the scale indicates that the individual's perception of SEM is at a good level.
Student Satisfaction and Self-Confidence in Learning Questionnaire | one month after intervention
  It evaluates student satisfaction and self-confidence in learning. The total number of items is 12. The scale is a 5-point Likert type and consists of the subscales "Satisfaction with Current Learning" and "Self-Confidence in Learning". The satisfaction with current learning subscale consists of 5 items, the self-confidence in learning subscale consists of 7 items, and there are no negative items. The sum of the subdimensions of the scale does not give the total score. Scale scores; It is obtained by dividing the sum of the sub-dimensions by the number of items. As the total score from the scale increases, student satisfaction and self-confidence in learning also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca çiçek okuyan, PhD, Principal Investigator — Manisa Celal Bayar University
Locations (2):
- Turkey (Türkiye) (2):
  - Manisa Celal Bayar University Faculty of Health Sciences, Department of Midwifery, Manisa
  - Yonca çiçek okuyan, Manisa